CLINICAL TRIAL: NCT05297838
Title: The Utilization of a Stationary Bike During Ice Bath While Using Virtual Reality (VR) to Determine Overall Pain Reduction
Brief Title: Stationary Bike Use During Ice Bath and Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Samuel Rodriguez, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 64860
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-08

CONDITIONS: Pain
Keywords: Ice bath; Virtual Reality; Stationary Bike
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ice Bath then VR and Bike During Ice Bath (Ice Bath vs VR Bike) (Active Comparator): Participants will immerse hand in ice bath and keep hand submerged as long as they can withstand the cold or until 4 minutes have elapsed, whichever comes first, while utilizing a VR headset. Participants will not be told of the specifics of the time limit, to avoid competitiveness and expectations and will be asked for pain scores every 30 seconds.
  After a washout period of 5 minutes, patients will immerse hand in ice bath keep hand submerged as long as they can withstand the cold or until 4 minutes have elapsed, whichever comes first, while utilizing a VR headset.Participants will not be told of the specifics of the time limit, to avoid competitiveness and expectations and will be asked for pain scores every 30 seconds.
  This occurred for both dominant and non-dominant hand. Randomization of dominant and non-dominant hands to the study conditions occurred prior to initiating the intervention.
  Interventions: Other: Stationary Bike; Other: Virtual Reality (VR) Headset; Other: Ice Bath
- VR with Ice Bath then Bike with VR During Ice Bath (VR vs VR Bike) (Active Comparator): Patients will immerse hand in ice bath keep hand submerged as long as they can withstand the cold or until 4 minutes have elapsed, whichever comes first, while utilizing a VR headset.Participants will not be told of the specifics of the time limit, to avoid competitiveness and expectations and will be asked for pain scores every 30 seconds.
  After a washout period of 5 minutes, Participants will immerse hand in ice bath while utilizing stationary bike and keep hand submerged as long as they can withstand the cold or until 4 minutes have elapsed, whichever comes first, while utilizing a VR headset. Participants will not be told of the specifics of the time limit, to avoid competitiveness and expectations and will be asked for pain scores every 30 seconds.
  This occurred for both dominant and non-dominant hand. Randomization of dominant and non-dominant hands to the study conditions occurred prior to initiating the intervention.
  Interventions: Other: Stationary Bike; Other: Virtual Reality (VR) Headset; Other: Ice Bath

INTERVENTIONS:
Other: Stationary Bike — Stationary Bike while hand is submerged in ice bath
Other: Virtual Reality (VR) Headset — VR headset containing gameplay
Other: Ice Bath — Pain was elicited via a cold pressor test, which is an established method of producing controlled and repeatable painful stimuli in an experimental setting

SUMMARY:
The purpose of this study is to evaluate the effectiveness of different technologies, in particular Virtual Reality, inclusive of passive content, active content, cognitive load modulation, and positive encouragement coaching to increase the pain threshold as assessed by immersing a hand in ice water while utilizing a stationary bike.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* English speaking
* Hearing intact

Exclusion Criteria:

* Patients who do not consent
* Are currently taking beta blockers or other chronotropic heart medication(s)
* Have a history of severe motion sickness
* Currently have nausea
* Currently experiencing seizures
* Are clinically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Self-Reported Pain Scores (Ice Bath vs VR Bike) | Duration of ice bath (approximately 0 - 4 minutes)
  Pain Scores will be collected during ice bath (maximum of 4 minutes) every 30 seconds via numeric rating scale (NRS), 0 being no pain, 10 being worst pain imaginable
Sympathetic Activation (VR vs VR Bike) | Duration of ice bath (approximately 0 - 4 minutes)
  Assessed via the electrodermal activity (EDA biosensor), which recorded skin conductance response density (SCRD) data in 30 second epochs. SCRD was recorded for the duration of the cold pressor test and one minute before and after submersion. The same primary and secondary outcome measures were collected at identical time points during the different cold pressor challenges on each hand

SECONDARY OUTCOMES:
Pain Tolerance (Ice Bath vs VR Bike) | Duration of ice bath (approximately 0 - 4 minutes)
  Defined by time of hand removal from the ice bath in seconds. 4 minute maximum.
Sympathetic Activation (Ice Bath vs VR Bike) | Duration of ice bath (approximately 0 - 4 minutes)
  Assessed via the electrodermal activity (EDA biosensor), which recorded skin conductance response density (SCRD) data in 30 second epochs. SCRD was recorded for the duration of the cold pressor test and one minute before and after submersion. The same primary and secondary outcome measures were collected at identical time points during the different cold pressor challenges on each hand.
Self-Reported Pain Scores (VR vs VR Bike) | Duration of ice bath (approximately 0 - 4 minutes)
  Pain Scores will be collected during ice bath (maximum of 4 minutes) every 30 seconds via numeric rating scale (NRS), 0 being no pain, 10 being worst pain imaginable and immediately after participant removed their hand from ice bath.
Pain Tolerance (VR vs VR Bike) | Duration of ice bath (approximately 0 - 4 minutes)
  Defined by time of hand removal from the ice bath in seconds. 4 minute maximum. The same outcome measure were collected at identical timepoints during both conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No